CLINICAL TRIAL: NCT03989128
Title: A Survey to Determine Cancer Patients' Perceptions of the Difficulties Encountered When Filling Opioid Prescriptions
Brief Title: Survey of Cancer Patients' Perceptions of Difficulties Encountered When Filling Opioid Prescriptions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0052; NCI-2019-02912 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0052 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Malignant Neoplasm; Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete a survey over 5-10 minutes
  Interventions: Other: Medical Chart Review; Other: Survey Administration

INTERVENTIONS:
Other: Medical Chart Review — Undergo medical chart review
  Other Names: Chart Review
Other: Survey Administration — Complete survey

SUMMARY:
This trial studies the problems that cancer patients face when filling prescriptions for opioids (medications that are used to manage pain). Pain is one of the most common symptoms among cancer patients. Opioid therapy is generally the treatment of choice for adequate management of cancer-related pain. Knowledge of these problems may help health care providers assess the most effective treatment options for cancer patients, and inform policy makers of the adjustments that need to be made to regulations to ensure cancer patients don't lose their access to opioids.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate patients' perceptions of overall difficulties when filling their opioid prescription.

SECONDARY OBJECTIVES:

I. To determine cancer patients' perceptions of financial, logistical, and psychosocial difficulties when filling their opioid prescription.

II. To evaluate the association between patient characteristics and patient difficulty filling opioid prescriptions.

OUTLINE:

Participants complete a survey over 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be on opioids provided by the Supportive Care Center (SCC), and must have visited the SCC 2 previous times for the purpose of opioid pain management. This will ensure that 1) patients will have been told that they are being prescribed an opioid as a treatment for pain, and 2) patients will have gone to a pharmacy to fill their opioid prescription a minimum of one time.
* Patients must be able to understand, read, write, and speak English.
* Patients must sign an informed consent document.
* Patients must have a cancer diagnosis.

Exclusion Criteria:

* Patients who have clinical evidence of cognitive impairment (Memorial Delirium Assessment Scale [MDAS] score of >= 13) as determined by the research staff, treating physician, or nurse.
* Patients who are considered to be in severe physical or emotional distress based on the assessment by the research staff.
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients on opioids for pain management provided by the Supportive Care Center
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Patients' perception of overall difficulties when filling opioid prescriptions | 2 years
  The proportion of patients who have experienced any difficulty when filling their prescription will be reported along 95% confidence intervals. Association of patients' characteristics with experiencing difficulty will be evaluated by Wilcoxon rank sum test and chi-square (Fisher's exact) test for continuous and categorical variables, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org